CLINICAL TRIAL: NCT01869933
Title: An Open Label Phase I Placebo Controlled, Dose Escalation Study Assessing the Ocular and Systemic Safety and Tolerability of OC-10X
Brief Title: Phase I Study Assessing the Ocular and Systemic Safety and Tolerability of OC-10X
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OcuCure Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OC-10X-102
Record Dates: First submitted 2013-05-28; First posted 2013-06-05 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Proliferative Diabetic Retinopathy (PDR)
Keywords: Proliferative, Diabetic, Retinopathy
MeSH Terms: conditions — Retinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1% OC-10X (Experimental): Subjects selected to Cohort I will receive active 1% OC-10X in OD (Oculus Dexter - right eye) and placebo (vehicle) in OS (Oculus Sinister - left eye) in the Period 1 dosing. On Study Day 1 the subjects will have a drop instilled in each eye by personnel at study hours 0, 3, 6 and 9, and be evaluated frequently throughout the day. Subjects will be examined on Study Day 2 (24 hours after first dose). On Study Day 3 (48 hours after the first dose), these subjects will commence Period 2 dosing, with the active (OD) or placebo (OS). Dosing will continue q.i.d. for an additional 13 days.
  Interventions: Drug: OC-10X
- 2% OC-10X (Experimental): Subjects selected to Cohort II will receive active 2% OC-10X in OD (Oculus Dexter - right eye) and placebo (vehicle) in OS (Oculus Sinister - left eye) in the Period 1 dosing. On Study Day 1 the subjects will have a drop instilled in each eye by personnel at study hours 0, 3, 6 and 9, and be evaluated frequently throughout the day. Subjects will be examined on Study Day 2 (24 hours after first dose). On Study Day 3 (48 hours after the first dose), these subjects will commence Period 2 dosing, with the active (OD) or placebo (OS). Dosing will continue q.i.d. for an additional 13 days.
  Interventions: Drug: OC-10X

INTERVENTIONS:
Drug: OC-10X

SUMMARY:
The present study is intended to evaluate the safety and tolerability of topical OC-10X Ophthalmic Suspension in healthy human subjects. OcuCure Therapeutics, Inc. (Roanoke, VA) has developed a lead compound, known as OC-10X, which is a selective tubulin inhibitor under development for the treatment of Proliferative Diabetic Retinopathy (PDR) and Age-related Macular Degeneration (AMD). When administered as a topical eye drop, OC-10X has demonstrated both anti-angiogenic (inhibition) and angiolytic (regression) properties in animal models of AMD. Unlike other therapies, OC-10X provides the efficacy of a vascular targeting agent without the traditional toxicity and works downstream independently of growth factors. As demonstrated by OcuCure's preclinical data, tubulin inhibition using OC-10X has promise as a new therapeutic approach. PDR is a major cause of blindness in adults and is also caused by the growth of abnormal blood vessels. These new blood vessels are fragile and may hemorrhage into the vitreous. PDR affects up to 80% of all diabetics who have had diabetes for 15 years or more. If administration of OC-10X is well tolerated as a topical eye drop and is well tolerated systemically, then OC-10X will have the potential to provide benefits to patients with ocular diseases associated with angiogenesis.

ELIGIBILITY:
Inclusion Criteria

1. Ability to provide approved written informed consent and comply with study-related procedures/assessments for the duration of the study, age > 18 years
2. Corrected visual acuity >20/25 in both eyes
3. IOP <21 mm Hg, with a difference between eyes of < 4 mm Hg
4. Ability to tolerate and self-administer vehicle eye drops.
5. Tolerance of a commercially available non-preserved, artificial tear solution
6. Normal slit lamp exam and dilated fundoscopic exam within one week previous to dosing
7. Normal clinical laboratory profiles for complete blood count, serum chemistry and electrolytes, and urinalysis with no clinically significant values
8. Be neither overweight nor underweight for his/her height as per BMI scale (18.5-24.9)
9. Female of childbearing potential:

   * Is practicing an acceptable method of birth control for the duration of the study, such as condoms, foams, jellies, diaphragm, IUD, or abstinence; or
   * Is postmenopausal for at least 1 year; or
   * Is surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy)

Exclusion Criteria

1. Evidence of organ dysfunction or any clinically significant deviation from the normal, in physical or clinical determinations
2. History of serious gastrointestinal, hepatic, renal, cardiovascular, pulmonary, neurological, hematological disease, diabetes, glaucoma, head-injury or coma
3. History of significant recurrent bacterial, viral or fungal infections
4. History of any psychiatric illness, which may impair the ability to provide written informed consent
5. Presence of disease markers of HIV 1 or 2, Hepatitis B or C viruses or syphilis infection
6. Presence of values which are significantly different from normal reference ranges and/or judged clinically significant for haemoglobin, total white blood cells count, differential white blood cell count or platelet count
7. Positive urinary screen testing of drugs of abuse (opiates, cannabinoids, amphetamines, barbiturates, benzodiazepines, cocaine)
8. Presence of values, which are significantly different from normal reference ranges and/or judged clinically significant for serum creatinine, blood urea nitrogen, serum aspartate aminotransferase, serum alanine aminotransferase, serum alkaline phosphatase, serum bilirubin, plasma glucose, serum cholesterol, serum electrolytes (sodium, potassium, chloride, calcium and phosphorus),serum proteins (albumin and globulin) and serum creatinine phosphokinase
9. Clinically abnormal chemical and microscopic examination of urine defined as presence of red blood cells, white blood cells (>4/High Power Field [HPF]), glucose (positive) or protein (positive)
10. Clinically abnormal electrocardiogram
11. Regular smokers, who smoke more than 10 cigarettes daily, or have difficulty abstaining from smoking
12. History of drug dependence or excessive alcohol intake on a habitual basis of more than 2 units of alcoholic beverages per day (1 unit equivalent to half pint of beer or 1 glass of wine or 1 measure of spirit) or have difficulty in abstaining from drinking
13. Subjects who, through completion of this study, would have donated and/or lost more than 400 mL of blood in past 2 months
14. History of ocular surgery, trauma, or chronic ocular disease
15. Current use of contact lenses or discontinuation of contact lens use within 2 weeks of the first dosing day
16. Any ocular abnormalities or ocular symptoms
17. Use of ocular agents (including eye drops) within the past 2 months or anticipated use of ocular agents during the study period
18. Systemic corticosteroid use within the past 6 months
19. History or evidence of ocular infection, inflammation, blepharitis, or conjunctivitis with 2 months; history of herpes simplex keratitis
20. Presence of a non-healing wound, ulcer, fracture, or any medical condition associated with bleeding.
21. Use of antimitotic or antimetabolite therapy within 2 months of enrollment.
22. Women who are pregnant or breastfeeding, or nonsterile or premenopausal women who refuse to use any form of contraception during and for at least 2 weeks following the final dose of study drug.
23. Enrollment in another investigational drug or device study within 2 months of study entry.
24. Known intolerance or hypersensitivity to any components/excipients in the study drug formulation.
25. Planned use during the study of any ocular or systemic medication, with the exception of oral contraceptives and short-term use of over-the-counter analgesics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Ocular Safety and Tolerability | 17 Days
  Ocular safety and tolerability will be assessed by subject query, biomicroscopy of anterior segment, ophthalmoscopy, measuring intraocular pressure (IOP) and checking visual acuity by modified Early Treatment Diabetic Retinopathy Study (ETDRS).

SECONDARY OUTCOMES:
Systemic Safety and Tolerability | 17 Days
  Systemic safety and tolerability will be examined by checking vital signs including heart rate, blood pressure, body temperature and respiratory rate, by electrocardiography (ECG) and performing a physical exam. Normal systemic function will be examined by routine blood draw for clinical chemistry, complete blood chemistry (CBC) and measure of plasma concentration of OC-10X.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Niaz Abdur-Rahman, MBBS,DO,MPH, Principal Investigator — Bangladesh Eye Hospital
Locations (1):
- Bangladesh Eye Hospital, Dhaka, Bangladesh